CLINICAL TRIAL: NCT03424447
Title: Stimulation of the Efferent Loop Before Loop Ileostomy Closure
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Basurto (Other)
Collaborators: Alberto Loizate Totoricaguena (Unknown); Pedro García Alonso (Unknown)
Responsible Party: Principal Investigator, ALBA VÁZQUEZ-MELERO, General Surgeon, Hospital de Basurto
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Hospital de Basurto
Record Dates: First submitted 2018-01-31; First posted 2018-02-07 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-01

CONDITIONS: Ileostomy - Stoma; Ileostomy; Complications; Stoma Ileostomy; Ileus Paralytic
MeSH Terms: conditions — Ileus

STUDY DESIGN:
Intervention Model Description: Ambispective cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non stimulated (No Intervention): Prospective data obtained from non stimulated patients
- Stimulated (Experimental): Prospective data obtaied from stimulated patients
  Interventions: Procedure: efferent limb stimulation

INTERVENTIONS:
Procedure: efferent limb stimulation
  Arms: Stimulated

SUMMARY:
The purpose of the study is to determine the impact of the efferent loop stimulation of a loop ileostomy prior to closure on postoperative complications such as ileus and hospital stay

DETAILED DESCRIPTION:
Stimulation was performed 3 weeks prior to the ileostomy closure using 500 cc of a thickening substance (saline and nutritional thickener) through the efferent limb.

ELIGIBILITY:
Inclusion Criteria:

* Patients with loop ileostomy
* Barium transit throught the efferent limb without leaks

Exclusion Criteria:

* Chemotherapy at the moment
* Ileostomy closure at the same admission than the ileostomy creation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2014-11-20; Primary Completion 2018-06-30 (Estimated); Study Completion 2018-10-30 (Estimated)

PRIMARY OUTCOMES:
postoperative ileus | during the admission for the ileostomy closure
  Need for a nasogastric tube
bowel movement | during the admission for the ileostomy closure
  day of hospital stay whe stool or flatus begins

SECONDARY OUTCOMES:
hospital stay | during the admission for the ileostomy closure
  days

CONTACTS AND LOCATIONS:
Overall Officials: Alba Vázquez-Melero, Principal Investigator — general surgeon
Locations (1):
- Hospital de Basurto, Bilbao, Vizcaya, Spain

IPD SHARING:
Plan to Share IPD: No